CLINICAL TRIAL: NCT05886725
Title: At-home Walking Cadence Functional Assessment and Recovery Trajectory for Older Adults Undergoing Major Surgery
Acronym: CADENCE
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB22-0556
Record Dates: First submitted 2022-12-06; First posted 2023-06-02 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Gait, Unsteady
Keywords: Walking Cadence; Surgery; Older Adult; Smartphone; Accelerometer; Recovery trajectory; Functional capacity; Activity; Major abdominal surgery
MeSH Terms: conditions — Gait Disorders, Neurologic; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Patients using Step Test Application and Accelerometer — Patients who are scheduled to have surgery at University of Chicago Medical Center (UCMC) who agree to use the step test application and study accelerometer before and after their surgery.

SUMMARY:
This is a prospective observational study looking at gait-cadence in older adults who are scheduled to have major abdominal surgery at the University of Chicago. The objective of the study is to evaluate whether gait-cadence, as measured from a patient's mobile device at-home, can provide an accurate assessment of a patient's functional status prior to major abdominal surgery and identify patients at risk of poor functional outcomes.

DETAILED DESCRIPTION:
Over 100,000 older adults undergo elective major abdominal surgeries in the US each year and many experience loss of mobility after surgery that requires post-acute care. Risk of mobility loss is greater for older adults unable to engage in moderate-intensity physical activity before surgery. Additionally, recovery trajectories to baseline mobility remains poorly understood for older adults and may impact readmission. Functional status assessment before surgery can identify interventions to help older adults improve walking capacity and improve recovery trajectories after surgery. However, almost no patients receive objective functional status tests before surgery due to logistical and practical barriers. Remote assessments performed independently by the patient using wearable technology, such as smartphones, may provide a solution. Smartphone accelerometers combined with open-source software can directly measure a patient's gait-cadence, or the number of steps taken per minute. This observational cohort of older adults undergoing major abdominal surgery will use a novel smartphone application to obtain remotely collected gait-cadence from usual and fast paced walks prior to their in-clinic visit. Investigators will then compare the at-home to the in-clinic usual and fast paced walks and measure their recovery trajectory after surgery through weekly at-home walks. Overall mobility will be assessed using ActiGraph accelerometers worn for a 7-day time period before and after surgery. The investigator's hypothesis is that gait-cadence measured during usual and fast pace walks at-home will 1) provide an accurate and easy to use functional assessment 2) identify patients at-risk of mobility loss and 3) determine walking recovery trajectories for older adults after surgery. Results from this study will provide important knowledge on mobility trajectories of older adults after major abdominal surgery and develop a novel approach to identify high-risk older adults. Further, this platform may be leveraged to deliver mobility interventions before surgery to improve patient outcomes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 60 years of age and scheduled for surgery.
* Access to a safe walking space roughly 30 ft in length. Safe walking spaces include a long hallway in the home, common use hallway in an apartment building or outside public area.
* Able to walk independently with or without an assistive device (e.g. cane or walker)

Exclusion Criteria:

* Inability to walk independently
* Surgery scheduled less than 7-days after APMC appointment
* Patients scheduled for orthopedic surgery
* Patients scheduled for neurological surgery
* Patients scheduled for cardiac surgery
* Non-English speaking.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are 60 years or older who have surgery scheduled at University of Chicago that can walk independently with or without an assistive device.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of gait-cadence measured from at-home and in-clinic walk tests as measured by ActivPAL accelerometers. | Baseline (Before surgery)
  ActivPAL accelerometer will be worn during in-clinic walk tests to serve as reference of steps walked during the at-home walk tests.

SECONDARY OUTCOMES:
Change in disability, as measured by the World Health Organization Disability Assessment Schedule (WHODAS) 2.0: 12-item. | Baseline (Before surgery), 1 month after surgery, 3 months after surgery
  The simple sum of the scores of the 12-items range from 0 to 48 with higher scores indicating greater disability.
Change in functional status, as measured by an interview in which participants will be asked, "At the present time, do you need help from another person to (complete the task)?" | Baseline (Before surgery), 1 month after surgery, 3 months after surgery
  Interview question will be asked for 13 different tasks. An increased need for personal assistance demonstrates greater functional status decline.
Change in global health, as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 - Global Health. | Baseline (Before surgery), 1 month after surgery, 3 months after surgery
  Total raw scores are between 4 and 20, and these can be converted to a T-score. Higher scores mean more of the concept being measured. For example, higher scores mean more health.
Change in pain interference, as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.1 - Pain Interference 6a. | Baseline (Before surgery), 1 month after surgery, 3 months after surgery
  Total raw score ranges from 6 to 30, and these can be converted to a T-score. Higher scores indicate greater pain interference on relevant aspects of a participant's life.
Change in gait-cadence after surgery | Weeks 1-8 after surgical procedure
  Gait-cadence will be measured at-home after surgery from weekly at-home walking tests from smartphone

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rubin, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No